CLINICAL TRIAL: NCT05196932
Title: A Pilot Study Investigating the Clinical Performance of a Novel, Point-of-care, Semi-quantitative Test for SARS-CoV-2 Antibodies in Patients Vaccinated Against COVID-19
Brief Title: COVID Card Pilot Study to Detect Antibodies to SARS-CoV-2
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Richard Gentry Wilkerson, Associate Professor, University of Maryland, Baltimore
Other Study IDs: HP-00099032
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID Card: Enrolled patients will receive antibody testing using both: 1) point-of-care, semi-quantitative SARS-CoV-2 antibodies test, 2) SARS-CoV-2 central laboratory antibodies test
  Interventions: Device: Novel point-of-care, semi-quantitative test for SARS-CoV-2 antibodies

INTERVENTIONS:
Device: Novel point-of-care, semi-quantitative test for SARS-CoV-2 antibodies — A drop of blood obtained by both finger-prick and venipuncture will be placed on the test card, which has been activated by the addition of diluent. Visual clumping of red blood cells (RBCs) will be seen within minutes if SARS-CoV-2 antibodies are present. Additionally, the COVID card is semi-quantitative, meaning that the yielded hemagglutination pattern will correlate with the concentration of antibodies in the serum.
  A research team member will be present at bedside to provide their interpretation based on an established visual agglutination scoring system.
  Other Names: Covid Card

SUMMARY:
This study aims to investigate the clinical performance characteristics of the novel point-of-care, semi-quantitative test for SARS-CoV-2 in the Emergency Department compared to the gold standard (ELISA).

DETAILED DESCRIPTION:
A prospective, non-blinded, non-randomized trial will be conducted at the Adult Emergency Department at the University of Maryland Medical Center and Adult Urgent Care Center, which is managed by the Department of Emergency Medicine, located in Baltimore, Maryland.

Patients meeting eligibility criteria and who have signed the research informed consent will be enrolled in this study. Subject data collected will include demographic information and past medical history. Upon enrollment into the study, a study team member will obtain a fingerstick blood sample and a sample of blood obtained during usual care venipuncture. Both fingerstick blood and blood from venipuncture will be run on the point-of-care, semi-quantitative test. The test should be expected to result within minutes after the blood sample is added to the agglutinin. An additional tube of blood will be obtained and sent to the local central laboratory for quantitative serum SARS-CoV-2 antibody testing.

Additional data will be collected on the reported or documented COVID-19 immunization status and reported or documented history of prior COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age > 18 years) emergency department patients
2. ED workup includes blood testing
3. Confirmed history of vaccination against SARS-CoV-2

Exclusion Criteria:

1. Known to be pregnant at the time of evaluation
2. Incarcerated at the time of evaluation
3. Requires the use of an interpreter
4. Patient is considered immunocompromised or has any other condition that the investigator feels makes the patient unsuitable for study inclusion.
5. Has any other condition that the investigator feels makes the patient unsuitable for study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient's presenting to the ED for symptoms other than Covid and are fully vaccinated (at least 2 vaccines). Patients with no suspicion of Covid symptoms or have tested negative.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Clinical Performance | 6 months
  To measure the diagnostic sensitivity, specificity, and accuracy compared to the gold standard central laboratory SARS-CoV-2 antibody test.

SECONDARY OUTCOMES:
Past Medical Conditions | 6 months
  To measure the diagnostic sensitivity, specificity, and accuracy compared to the gold standard central laboratory SARS-CoV-2 antibody test relative to patient past medical conditions
Time Since Vaccination | 6 months
  To measure the diagnostic sensitivity, specificity, and accuracy compared to the gold standard central laboratory SARS-CoV-2 antibody test relative to the time since vaccination
Inter-Rater Reliability | 6 months
  To measure differences in interpretation (scoring) of hemagglutination patterns between study team members.
Type of Blood | 6 months
  The test characteristics of blood obtained by fingerstick will be compared to that of blood obtained by venipuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Wilkerson, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Systems, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IDP will not be made available to other researchers.

REFERENCES:
- [Background] Kruse RL, Huang Y, Lee A, Zhu X, Shrestha R, Laeyendecker O, Littlefield K, Pekosz A, Bloch EM, Tobian AAR, Wang ZZ. A Hemagglutination-Based Semiquantitative Test for Point-of-Care Determination of SARS-CoV-2 Antibody Levels. J Clin Microbiol. 2021 Nov 18;59(12):e0118621. doi: 10.1128/JCM.01186-21. Epub 2021 Sep 1. PMID 34469185